CLINICAL TRIAL: NCT02127411
Title: Adaptation and Evaluation of the Mindfulness-Based Relapse Prevention Program for Cessation and/or Reduction of Benzodiazepine Chronic Use to Induce Sleep Among Women
Brief Title: Effectiveness of Mindfulness Based Relapse Prevention for Chronic Users of Benzodiazepines
Acronym: MBRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Ana Regina Noto, Adjunct Professor at the Psychobiology Department, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MBRP BZD; CNPq and Fapesp (Other Grant/Funding Number: CNPq Decit 07/2013; CNPq FAPs 71/2013; FAPESP 2013/20367-6)
Record Dates: First submitted 2014-03-10; First posted 2014-04-30 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Benzodiazepine Dependence
Keywords: Mindfulness; Benzodiazepines; Sleep; Dependence; Relapse Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness-based relapse prevention (Experimental): Mindfulness-Based Relapse Prevention
  Interventions: Behavioral: Mindfulness-Based Relapse Prevention
- Waitlist (No Intervention): this group will stay in the waitlist until the end of follow-up assessments, when they will receive the intervention

INTERVENTIONS:
Behavioral: Mindfulness-Based Relapse Prevention — The MBRP is an adjuvant treatment for people that have been treated for drug use related problems
  Arms: Mindfulness-based relapse prevention

SUMMARY:
Benzodiazepines (BZD) are the most prescribed psychiatric drugs in Brazil, especially for women. Although it is recommended that the use of BZD is not greater than four weeks, there are many cases of prolonged use due to the lack of treatment options for dealing with complaints of insomnia. Given this, the aim of this project is to evaluate the program Mindfulness-Based Relapse Prevention (MBRP) for adult women with chronic use of benzodiazepine (BZD) to induce sleep. Specifically aims to evaluate if the MBRP program, can reduce the pattern of use and level of dependence of chronic users of BZD under gradual reduction (tapering) or cessation of the use of BZD. This study will be conducted at the Drug Dependency Unit (UDED) of the Department of Psychobiology of Federal University of São Paulo. The study will count with two groups: intervention group (IG) and control group (CG) (that will stay in the waitlist until the eighth month . The sample will comprise 100 women with chronic use of BZD as hypnotics, 50 will be randomized in the IG condition and 50 in the CG condition. Changes will be evaluated on several variables such as cessation and dependence of BZD, quality of life, sleep, anxiety, depression and sexual satisfaction before and after the intervention in both groups. The data will be submitted to descriptive and inferential bivariate and multivariate statistic analyzes. It is hoped that this study create subsidies for the development of complementary interventions for the management of withdrawal symptoms in chronic users of BZD.

ELIGIBILITY:
Inclusion Criteria:

* Literate adult women
* Using benzodiazepine (BZD) for inducing sleep for at least 03 months (90 days), for at least four times a week.

Exclusion Criteria:

* Having practiced regularly meditation, yoga or similar previously, at least once a week, for at least three months, or have carried this practice regularly at least once a week in the last year for at least one month
* Neurological disorders, anxiety refractory to other treatments or insomnia secondary to other severe clinical conditions, which the BZD withdrawal is considered as a potential risk for worsening
* Presence of not controlled clinical disease or of greater severity, such as cancer, schizophrenia, epilepsy
* Presence of psychiatric illness which withdrawal of BZD is considered a potential risk for worsening
* Dependence or abuse of alcohol or other drugs, except tobacco
* In acute treatment for psychological or psychiatric problems
* Be participating in a tapering BZD protocol, or similar

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
reduction of benzodiazepine use | Change from baseline in benzodiazepine use at 8 months.
  We will evaluate the reduction through a percentual comparison between the dose the patient is using at follow-up assessments and the dose related at the beginning of the study.
Severity of insomnia | Change from baseline in insomnia severity at 8 months
  We will evluate the severity os insomnia with the Insomnia Severity Index (ISI) which is a self-report questionnaire and consists of seven items that evaluate severity of sleep onset, sleep maintenance and early morning awakening problems; sleep dissatisfaction; interference of sleep difficulties with daytime functioning; noticeability of sleep problems by others, and distress caused by sleep difficulties. The score for each item ranges from 0 to 4, totaling 0 to 28 points, with a higher score indicating greater insomnia severity.

SECONDARY OUTCOMES:
Stage of change related to benzodiazepine use | Change from Baseline of the stage of change at 8 months
  This will be measured by an analogic rule from 1 to 10, in which 1 means "not ready to change" and 10 means "actively working in the change"
self report mindfulness level | Change in mindfulness level from baseline at 8 months
  This will be measured with the self report questionnaires: Five Facet Mindfulness Questionnaire. This is a self-report questionnaire and do not have a specific metric to measure mindfulness. The scores are absolute and a higher score denotes higher levels of mindfulness
Level of Benzodiazepine dependence (from mild to severe) | change in benzodiazepine dependence severity from baseline at 8 months
  this will be measured through the Benzodiazepine Dependence Self-Report Questionnaire, which is a self report questionnaire and do not provides a specific metric to measure the severity of dependence.
Symptoms of depression | Change in symptoms of depression from baseline at 8 months
  The symptoms of depression will be measured through the Center for Epidemiologic Studies Depression Scale - CES-D. As it is a self report scale, there is no specific metric to measure depression.
Sleep Quality | Change in sleep quality from baseline at 8 months
  will be measured through the Pittsburgh Sleep Quality Index
menopausal symptoms (Kupperman index) | change in menopausal symptoms from baseline at 8 months
Female Sexual Satisfaction | change in female sexual satisfaction from baseline at 8 months
presence of benzodiazepines metabolites identified with a toxicology urinalysis | Change in benzodiazepine metabolites from baseline at eight months
Epigenetic modifications | Baseline and 2 month follow-up
  Blood collection will be held, and the plasma will be analyzed to evaluate levels of homocysteine and cysteine , two aminoacids that are related to epigenetic modifications that can modulate the behavioral responses resulting from the practice of meditation
Trait Anxiety | Baseline, 2, 4 6 and 8 months follow-ups
  Evaluated using the State and Trait Anxiety Index (STAI), validated in Brazil (α = 0.87). We used only the subscale of trait anxiety, less susceptible to environmental alterations. This subscale is composed by 20 items on a four-point Likert scale ("almost never", "sometimes", "often", "almost always"), in which the participant is instructed to answer "how do you usually feel". The Cronbach α in this sample was 0.90.

CONTACTS AND LOCATIONS:
Overall Officials: Ana R Noto, PhD, Study Chair — Affiliate Professor
Locations (1):
- Drug Dependency Unit of the Universidade Federal de São Paulo (UDED), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Barros VV, Opaleye ES, Demarzo M, Curado DF, Bowen S, Hachul H, Noto AR. Effects of Mindfulness-Based Relapse Prevention on the Chronic use of Hypnotics in Treatment-Seeking Women with Insomnia: a Randomized Controlled Trial. Int J Behav Med. 2022 Jun;29(3):266-277. doi: 10.1007/s12529-021-10002-4. Epub 2021 May 19. PMID 34013489